CLINICAL TRIAL: NCT01846546
Title: Dynamic Changes of Cerebrospinal Fluid Endostatin Concentrations in Patients With Severe Traumatic Brain Injury.
Brief Title: Cerebrospinal Fluid Endostatin/Collagen XVIII Concentrations in Patients With Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Other Study IDs: ES-TBI 10JC
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury;; Endostatin/collagen XVIII;; Cerebrospinal fluid;; Prognosis
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Traumatic Brain Injury: Patients with severe TBI (Glasgow Coma Scale GCS score of 8 or less) requiring continuous lumbar drainage of CSF

SUMMARY:
Angiogenesis is an important pathophysiological response to traumatic brain injury (TBI) and modulated by pro- and anti-angiogenic factors. Recent studies have suggested that endogenous angiogenesis inhibitor endostatin/collagen XVIII might play an important role in the secondary brain injury following TBI. The aim of this study was to investigate early changes in the concentrations of CSF endostatin/collagen XVIII after TBI and evaluated the relations of endostatin/collagen XVIII to injury severity and clinical outcome. Endostatin/collagen XVIII concentrations were measured serially for 1 week after hospitalization by using the enzyme linked immunosorbent assay method in the cerebrospinal fluid of 30 patients with TBI and a Glasgow Coma Scale score of 8 or less on admission. Comparative analysis were used to determine if its serial changes correlate with the GCS score and prognosis. Receiver operating characteristic curve was used to appraise the value of CSF endostatin/collagen XVIII levels in predicting the prognosis of patients with severe head injury.

DETAILED DESCRIPTION:
Patients with severe TBI (Glasgow Coma Scale score of 8 or less) requiring continuous lumbar drainage of CSF were included in the study. Patients delivered within 4 h whose highest abbreviated injury score was 3 or less (other than head injury) were considered to be isolated TBI cases and were included. To avoid interfering factors, patients who suffered open or combined injuries, had existing prior neurological disease were excluded. Those who died within the first week of hospitalization and/or whose serial cerebrospinal fluid samples could not be obtained were also excluded as having incomplete data. Accordingly, 30 patients were analyzed in this study. Demographic data, including age, gender, mechanism of trauma and GCS score at admission were documented when the patients arrived at the emergency room. The control group comprised 20 patients whose cerebrospinal fluid was examined via lumbar puncture for investigation of suspected neurological disease. All patients had normal neurological examination, negative imaging studies, and none had evidence of trauma or preexisting neurological disease, including tumors, vascular anomalies, or abnormalities of cerebrospinal fluid. The study had approval from the hospital ethics committee and informed consent for participating in the study was obtained from an appropriate member of each patient's family before performance of lumbar drainage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe TBI (GCS score of 8 or less) requiring continuous lumbar drainage of CSF. Patients delivered within 4 h whose highest abbreviated injury score (AIS) was 3 or less (other than head injury) were considered to be isolated TBI cases and were included.

Exclusion Criteria: Patients who suffered open or combined injuries, had existing prior neurological disease were excluded. Those who died within the first week of hospitalization and/or whose serial CSF samples could not be obtained were also excluded as having incomplete data.

-

Ages: 16 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Of the 30 patients with severe TBI, twenty were male and ten were female. The patients' age ranged from 16 to 82 years, with mean age of 51.1 years. The mechanisms of trauma included motor vehicle collisions, falls, heavy strikes (patients who were hit by heavy objects such as bricks, sticks, or falling objects) and assaults. Types of lesions, as evidenced by radiologic and neurologic symptoms or signs, included cerebral contusions/lacerations, intracranial hematomas, brain stem injury and diffuse axonal injury.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Enzyme-linked immunosorbent assay | 6 months
  This assay employs the quantitative sandwich enzyme immunoassay technique. In brief, a monoclonal antibody specific for endostatin/collagen XVIII had been pre-coated onto a microplate.

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Li Tian, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

REFERENCES:
- [Derived] Chen H, Xue LX, Cao HL, Chen SW, Guo Y, Gao WW, Ju SM, Tian HL. Endostatin/collagen XVIII is increased in cerebrospinal fluid after severe traumatic brain injury. Biomed Res Int. 2013;2013:402375. doi: 10.1155/2013/402375. Epub 2013 Sep 8. PMID 24089677